CLINICAL TRIAL: NCT04589182
Title: Assessing the Symptomatic Benefit of Acoustic Slow Wave Enhancement in Parkinson Disease: A Randomized, Double-Blind and Placebo-Controlled Crossover Study
Brief Title: Assessing the Symptomatic Benefit of Acoustic Slow Wave Enhancement in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian Baumann (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor-Investigator, Christian Baumann, Professor, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PDSL-EDS
Record Dates: First submitted 2020-09-29; First posted 2020-10-19 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment; Huntington Disease
Keywords: sleep; neurodegeneration; slow- wave sleep
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Huntington Disease; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, sham-controlled cross-over trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: During data collection, patients will be blinded to the condition. The leading experimenter will be unblind and have access to the keys that define whether the interventions, namely intervention 1 and intervention 2, are sham or verum. However, all experimenters will be blinded for analysis of outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Patients will receive all-night auditory stimulation during sleep over 3 nights using a portable, safe, in-home device (MSHL-SleepBand). This device records biosignals (EEG) and precisely plays tones (between 45-65 dB, maximum 80 dB) targetted to the up-phase of sleep slow waves.
  Interventions: Device: MHSL- SleepBand
- Sham (Sham Comparator): Patients will receive all-night sham stimulation over 3 nights, i.e. the wearable stimulation device will be applied (EEG will be recorded), but no tones will be played.
  Interventions: Device: Sham

INTERVENTIONS:
Device: MHSL- SleepBand — The MHSL-SleepBand (sleep headband) is easy to apply and only involves attachment of sticky electrodes on different locations on the face/behind ear to be able to measure EEG (electroencephalogram), EOG (electrooculogram) and EMG (electromyogram). Brief tones at a low volume (around 60 dB, comparable to conversation) will be applied, when slow waves are present in the course of the sleep period and other criteria are fulfilled. Auditory stimulation will start with a specific volume that has been adjusted to the individual hearing capacity (usually between 45-65 dB; maximum 80 dB). The stimulation is performed in a way that the general structure of sleep (e.g. duration, sleep cycling, etc.) is unchanged.
  Other Names: Auditory SWS stimulation
  Arms: Verum
Device: Sham — Playing no tones during non- Rapid Eye Movement (NREM) sleep but wearing the device and recording the biosignals over a period of 3 nights, every night.
  Other Names: Sham stimulation
  Arms: Sham

SUMMARY:
The study is a randomized, double-blind, sham-controlled cross-over trial to assess the efficacy as well as safety and tolerability of auditory SWS enhancement on measured outcomes in Parkinson disease (PD) patients with disturbed nighttime sleep.

Additionally, the investigators will assess the feasibility and efficacy of auditory slow-wave sleep (SWS) enhancement in Mild Cognitive Impairment (MCI) and Huntington Disease (HD) patients in a pilot study.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, sham-controlled cross-over trial to assess the efficacy as well as safety and tolerability of auditory SWS enhancement on measured outcomes in PD patients with disturbed nighttime sleep. Patients will be randomized to 2 groups: Group 1 will first be treated with auditory stimulation for 3 nights and then - after a wash-out period of 4 nights - switched to 3 nights of sham stimulation. Group 2 will first receive sham-stimulation for 3 nights and then switch to 3 nights of auditory stimulation treatment. The wash-out period in between will be 4 nights. Patients and investigators assessing the outcomes will be blinded to the conditions. All interventions will take place at the patients' homes.

The pilot study is aimed at assessment of safety, tolerability, feasibility and efficacy of auditory SWS enhancement on measured outcomes in MCI and HD patients with disturbed nighttime sleep. Patients will be treated with verum or sham auditory stimulation for 2 consecutive nights. All interventions will take place at the patients' homes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Diagnosis of PD along international criteria with mild to moderate disease severity (Hoehn- Yahr (HY) stages ll-lll),
* Self-reported sleep problems and subjectively impaired sleep quality (PDSS-2 sleep quality subscale (items 1-3 and 14) ≥7)
* Stable home situation (e.g. long-term place to live) that allows for reliable application of intervention for the duration of the study
* Ability to apply the intervention for the duration of study, either alone or with help of co-habitant
* Sufficient German language comprehension to follow the study procedures and answer all questions related to the study outcomes
* Dosing of dopaminergic and other PD treatment must have been stable for at least 14 days prior to the first intervention period
* Negative pregnancy test during screening (except in women who are surgically sterilized/hysterectomized or post-menopausal for longer than 1 year),
* Age above 18 years

Exclusion Criteria:

* Known presence of neurologic (other than PD), psychiatric, or sleep disorders (others than associated with PD)
* Parkinsonism without response to levodopa; Atypical Parkinsonian syndromes
* Severe medical conditions as renal insufficiency, liver failure or congestive heart failure
* The regular use of benzodiazepines and other central nervous system (CNS)-depressant substances, as well as melatonin and other sleep inducing substances
* Inability to hear the tones produced by the MHSL-SleepBand device
* Absence of slow-wave enhancement by auditory stimulation during the screening night
* Skin disorders/problems/allergies in face/ear area that could worsen with electrode application
* Failure to give informed consent
* Known or suspected drug- or medication abuse
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, cognitive deficits
* Cognitive impairment (Montreal Cognitive Assessment - MoCA <24)
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment in the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Shift work (work during the night)
* Travelling more than 2 time zones in the last month before intervention starts or during intervention (start of intervention will be adapted to fit with this criteria)
* Substance or alcohol abuse (i.e. > 0.5 l wine or 1 l beer per day)
* High caffeine consumption (> 5 servings/day; including coffee, energy drink)
* Planned medical intervention of substantial relevance, e.g. surgery, during intervention (routine assessments, e.g. check-ups will be allowed)
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female patients of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Please note that female patients who are surgically sterilized/hysterectomized or postmenopausal for longer than 1 year are not considered as being of child bearing potential.

Pilot studies:

Inclusion criteria:

* Informed Consent as documented by signature (see Informed Consent Form),
* Age above 18 years
* The diagnosis of MCI along international criteria or manifest HD (diagnosis of HD confirmed by genetic testing, patients above the age of 18 years, manifest HD, diagnostic confidence of 4)
* Stable home situation (e.g. long-term place to live) that allows for reliable application of intervention for the duration of the study,
* Stable regimen of therapeutic drugs for at least 2 weeks prior to the intervention,
* For HD patients: self-ambulatory
* Native German speaker or good understanding of German. Translation assistance will be accepted, if this will allow a nonnative German speaker to comprehensively follow the study protocol including all questionnaires
* Ability to apply the intervention for the duration of study, either alone or with help of co-habitant.

Exclusion criteria:

* MCI: Present diagnosis of neurologic (other than MCI), interfering psychiatric, or severe internal disease
* HD: Diagnosis of juvenile onset HD
* HD: History of co-morbid neurological conditions (e.g. multiple sclerosis or stroke), interfering psychiatric or cognitive disorders
* Severe medical conditions, such as renal insufficiency, liver failure or congestive heart failure
* Inability to hear the tones to be applied during sleep when awake
* Skin disorders/problems/allergies in face/ear area that could worsen with electrode application
* MCI: absence of a cohabitant who could assist with study applications and procedures
* Failure to give informed consent
* Known or suspected drug- or medication abuse
* Inability to follow the procedures of the study, e.g. due to language problems, cognitive deficits,
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* substance or alcohol abuse (i.e. > 0.5 l wine or 1 l beer per day),
* Planned medical intervention of substantial relevance, e.g. surgery, during intervention (routine assessments, e.g. check-ups will be allowed)
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female patients of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Please note that female patients who are surgically sterilized/hysterectomized or post-menopausal for longer than 1 year are not considered as being of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality | assessed before and after each intervention (day 1 and 4, day 7 and 10)
  Changes in subjective sleep quality measured with adapted version of Parkinson Disease Sleep Scale (PDSS2), questions on a scale of 0-4, with 0 indicating better sleep
Pilot study: feasibility of acoustic SWS enhancement | assessed after intervention (day 10)
  Feasibility of acoustic SWS enhancement in MCI and HD patients (enhancement of slow-waves measured with EEG)

SECONDARY OUTCOMES:
Vigilance | assessed before and after each intervention (day 1 and 4, day 7 and 10)
  Changes in vigilance measured using Psychomotor Vigilance Test (PVT)
Sleep benefit on motor performance | assessed before and after each intervention (day 1 and 4, day 7 and 10)
  Changes in motor performance assessed with focus motor assessment
Momentary sleepiness | assessed before and after each intervention, and every morning and evening during the intervention (day 1 until 4, day 7 until 10)
  Changes in momentary sleepiness assessed with Karolinska Sleepiness Scale (KSS) on a scale 1-10, with 1 indicating extreme alertness and 10 indicating extreme sleepiness
Average sleepiness | assessed every evening during the intervention (day 1 until 4, day 7 until 10)
  Average sleepiness throughout the day measured with VAS on a scale 0-100, with 100 indicating extreme sleepiness
Mood | assessed every evening during the intervention (day 1 until 4, day 7 until 10)
  Changes in mood assessed with Visual Analog Scale (VAS) on a scale 0-100, with 100 indicating extremely good mood
Restorative effect of sleep | assessed every morning during the intervention (day 1 until 4, day 7 until 10)
  Changes in restorative effect of sleep using VAS, on a scale 0-100, with 100 indicating very refreshing sleep
Slow wave enhancement | assessed every night of the intervention (day 1 until 4, day 7 until 10)
  Enhancement of slow waves with auditory stimulation, measured with EEG
Auditory stimulation algorithm performance | assessed every night of the intervention (day 1 until 4, day 7 until 10)
  Performance of algorithm detecting and stimulating slow waves, measured with EEG
Pilot study: changes in mood | before and after intervention (day 1 and 4, day 7 and 10)
  changes in mood assessed on VAS (Visual Analog Scale) on a scale 0-100, with 100 indicating extremely good mood
Pilot study: changes in sleep quality | before and after intervention (day 1 and 4, day 7 and 10)
  changes in sleep quality assessed on VAS (Visual Analog Scale) on a scale 0-100, with 100 indicating extremely good sleep quality
Pilot study: changes in sleepiness | before and after intervention (day 1 and 4, day 7 and 10)
  changes in sleepiness assessed on VAS (Visual Analog Scale) on a scale 0-100, with 100 indicating extreme sleepiness

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Neurology department, Zurich, Canton of Zurich, Switzerland